CLINICAL TRIAL: NCT06855472
Title: Comparison of the MAR Method and the Visual Estimation Method in Predicting External Blood Loss in Health Students
Brief Title: The MAR Method Versus the Visual Estimation Method in Predicting External Blood Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Betül Akbuğa Özel (Other)
Collaborators: Baskent University (Other)
Responsible Party: Sponsor-Investigator, Betül Akbuğa Özel, Assistant Professor, MD, FTBEM, MSc, PhD, Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KA17/92
Record Dates: First submitted 2025-02-18; First posted 2025-03-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Blood Loss
Keywords: blood loss; clinical skills; emergency medicine; medical students; paramedics; randomized controlled trial; simulation training
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Our study does not involve treatment, prevention, diagnosis, supportive care, screening, or medical devices. Instead, it is a randomized controlled trial that focuses on clinical skills training for estimating external blood loss in emergency medicine. The study designed a monocenter, double-blind, randomized, parallel-group, and controlled clinical educational study.
Who Masked: Participant, Investigator
Masking Description: Participant: Second-year paramedic student or second-year medical student, having received no theoretical or practical training in predicting external blood loss (N:237) Investigator: Student, provided planned training to participants, recorded outcome parameters Researcher: faculty member, prepared three different simulated environments and scenarios, provided planned training to investigators, oversaw flow of participants across study arms and recorded outcome parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Visual Estimation Method (Control), (n1:70) (No Intervention): The Visual Estimation Method is the most commonly used technique for estimating external blood loss. It relies on quick visual assessment rather than precise measurement, providing an estimate within seconds.
- Group 2: The MAR Method (Intervention), (n2:70) (Experimental): The MAR (Merlin, Alter, Raffel) method, which was first described by Merlin et al. in 2009, is an alternative clinical skill recommended for estimating the amount of external blood loss on flat surfaces and does not depend on visualization. The method can learn within 1-2 minutes. In this method, the participants are given 60 sec to complete their estimations.
  Interventions: Other: The MAR method

INTERVENTIONS:
Other: The MAR method — The study was conducted in three isolated stations. Two faculty researchers designed the scenarios, while three others supervised training. Medical student investigators recorded blood loss estimates and estimation times.
  Before the study, investigators received 20-minute training. Participants and investigators were blinded to actual blood volumes. Group 1 and Group 2 attended a 10-minute briefing, including consent and study introduction.
  The study had two phases. In Phase 1, Group 1 used the Visual Estimation (VE) method, while Group 2 received a 2-minute MAR method training before making estimations. In Phase 2, Group 1 was trained in the MAR method and repeated estimations.A data form recorded demographics, blood loss estimates, and estimation times.
  Group 1's VE data and Group 2's MAR data were compared between groups, while Group 1's VE and MAR data were analyzed within the group. Combined MAR data from both groups were used to assess the impact of gender, height, and weight.
  Arms: Group 2: The MAR Method (Intervention), (n2:70)

SUMMARY:
The goal of this educational clinical trial is to determine whether the MAR method is more effective than the Visual Estimation method for estimating blood loss. It also aims to assess whether factors such as gender, weight, and height influence blood loss estimates when using the MAR method.

The main research questions it aims to answer are:

* Does the MAR method provide more accurate blood loss estimates than the Visual Estimation method on flat, non-absorbent surfaces?
* Does the MAR method take longer to estimate blood loss compared to the Visual Estimation method?
* Do demographic factors such as gender, height, and weight affect blood loss estimates using the MAR method?
* Do these demographic factors also influence the time required for estimation using the MAR method? Researchers will compare the MAR method with the Visual Estimation method to determine whether the MAR method is a useful tool for accurately estimating external blood loss in clinical skill training.

Participants will:

* Sign an Informed Consent Form at the start of the study
* Receive a 10-minute orientation session
* Receive a 2-minute MAR method training (for the intervention group-)
* Use either the MAR method or the Visual Estimation method for up to 60 seconds at each of the three stations
* Receive a 2-minute MAR method training (for the control group)
* Use the MAR method for up to 60 seconds at each of the three stations (for the control group)

DETAILED DESCRIPTION:
Preliminary Preparation:

For this study, the Professional Skills Laboratories were used as the physical setting. The scenarios were set up at three different stations, each positioned in a separate corner of a large room. Room dividers separated the stations, and each had a designated entrance and exit to prevent participants who had completed their estimations from encountering those who had not yet participated.

Two researchers designed three distinct simulated environments and scenarios for the study. A synthetic blood product was used to enhance the realism of the simulated blood loss cases. In line with the MAR method's design principles, all three stations featured flat, non-absorbent surfaces.

* Station 1: An acrylic (plexiglass) surface with 75 ml of blood.
* Station 2: A flat, varnished wood surface with 150 ml of blood.
* Station 3: A vinyl surface with 750 ml of blood.

Research Staff:

Three faculty researchers were present in the simulation area, overseeing orientation training for investigators and participants and coordinating activities at each station. Additionally, three medical student investigators were assigned to record blood volume estimates and estimation times.

Randomization:

Out of 237 eligible participants, 140 met the inclusion criteria and consented to participate. Since students from both departments had similar academic levels, ages, educational backgrounds, and no prior formal training in external blood loss estimation, the researchers used a non-stratified selection method. Participants were randomly assigned into two equal groups of 70 using a block randomization method (1:1 ratio) via the online service https://researchrandomizer.com/.

To assign participants, group names were written on paper, placed in a bag, and selected blindly.

* Group 1: Control group (Visual Estimation method), (n1:70).
* Group 2: Experimental group (MAR method), (n2:70). Group assignments were revealed to participants only when they arrived at the simulation room. To ensure allocation concealment, an independent researcher conducted both the randomization and group assignment before the trial began. While faculty researchers who prepared the stations knew the actual blood volumes, participants and study investigators who recorded the data were blinded to this information.

Study Description:

Student investigators at the stations received a 20-minute orientation before the study, covering its purpose, workflow, data form usage, and chronometer operation. Investigators recorded data in real-time as estimations were made. Neither participants nor investigators knew the actual blood volumes at the stations (double-blind design). At the start of the study, both groups received a 10-minute briefing, including:

* Signing the consent form
* Explaining the study's purpose
* Introducing the simulation lab and research team

To clearly describe the procedures, the study is presented in two distinct periods. Period I was conducted to obtain the primary outcomes based on the primary objectives of the study. During this period::

* Group 1 (Control): Estimated blood loss using the Visual Estimation (VE) method.
* Group 2 (Experimental): Received 1-2 minutes of MAR method training separately, then estimated blood loss using the MAR method at all three stations.

Investigators at each station recorded blood volume estimates and estimation times for both groups. Researcher analysed data providing intergroup records (Visual estimation method [n1] vs MAR method [n2]) and intragroup records (Visual method [n1] vs MAR method [n1])

Period II process was conducted to obtain the secondary outcomes based on the secondary objectives of the study. In this period::

•Group 1 (Previously Control): Received 1-2 minutes of MAR method training separately, then estimated blood loss using the MAR method at all three stations.

Investigators recorded blood volume estimates and estimation times. For secondary outcomes, data from 140 participants (MAR method [n2] plus MAR method [n1]) were analyzed to determine whether gender, height, and weight influenced blood loss estimates and estimation durations using the MAR method.

ELIGIBILITY:
Inclusion Criteria:

* Being a second-year paramedic or medical student
* No prior theoretical or practical training in estimating external blood loss
* Willingness to participate in the study

Exclusion Criteria:

* Not being a second-year paramedic or medical student
* Having received theoretical or practical training in estimating external blood loss
* Declining to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Blood loss volume estimate | From enrollment to the completion of method application in 20 minutes.
  Blood loss volume estimates using the MAR and Visual Estimation (VE) methods were recorded in milliliters (ml). The participants had 60 seconds to complete their estimations at each station. Participants' verbal estimates were documented by researchers at each station on the study record form. Blood loss volume estimates obtained using Group 1's VE method (n1:70) Group 2's MAR method (n2:70) were compared between the groups. Blood loss volume estimates obtained using Group 1's VE method and MAR method (n1:70) were then compared within the group.
Blood loss estimation time | From enrollment to the completion of method application in 20 minutes.
  The blood loss estimation times for the MAR and VE methods were recorded in seconds. The participants had 60 seconds to complete their estimations at each station. A chronometer was used for each measurement. Blood loss estimation times obtained using Group 1's VE method (n1:70) and Group 2's MAR method (n2:70) were compared between the groups. Blood loss estimation times obtained using Group 1's VE method and MAR method (n1:70) were then compared within the group.

SECONDARY OUTCOMES:
Blood loss volume estimate of each participant using the MAR method | From enrollment to the completion of method application in 25 minutes.
  In Phase 1, data from Group 2's MAR application (n2:70) and in Phase 2, data from Group 1's MAR application (n1:70) were combined, resulting in a total of 140 data points (n1:70 + n2:70). The analysis examined the relationship between blood loss estimates and participants' gender, height, and weight.
Blood loss estimation time of each participant using the MAR method | From enrollment to the completion of method application in 25 minutes.
  In Phase 1, data from Group 2's MAR application (n2:70) and in Phase 2, data from Group 1's MAR application (n1:70) were combined, resulting in a total of 140 data points (n1:70 + n2:70).The analysis examined the relationship between blood loss estimation times and participants' gender, height, and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Akbuga Ozel, Asst.Prof., Principal Investigator — Ankara Yıldırım Beyazıt University, Faculty of Medicine, Ankara Bilkent City Hospital, Department of Emergency Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Baskent University, Ankara, Ankara
  - Ankara Yıldırım Beyazıt University, Faculty of Medicine, Ankara Bilkent City Hospital, Department of Emergency Medicine, Ankara, Ankara

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available. The IPD belongs to Baskent University; therefore, this decision must be made at the institutional level.

REFERENCES:
- [Background] Merlin MA, Alter SM, Raffel B, Pryor PW 2nd. External blood loss estimation using the MAR Method. Am J Emerg Med. 2009 Nov;27(9):1085-90. doi: 10.1016/j.ajem.2008.07.039. PMID 19931755
- [Background] Yeung CY, Yim WW, Chan SY, Lo RSL, Leung LY, Hung KKC, Graham CA. Improvement of blood loss volume estimation by paramedics using a pictorial nomogram: A developmental study. Injury. 2017 Dec;48(12):2693-2698. doi: 10.1016/j.injury.2017.10.045. Epub 2017 Oct 31. PMID 29108791
- [Background] Ashburn JC, Harrison T, Ham JJ, Strote J. Emergency physician estimation of blood loss. West J Emerg Med. 2012 Sep;13(4):376-9. doi: 10.5811/westjem.2011.9.6669. PMID 22942938
- [Background] Williams B, Boyle M. Estimation of external blood loss by paramedics: is there any point? Prehosp Disaster Med. 2007 Nov-Dec;22(6):502-6. doi: 10.1017/s1049023x0000532x. PMID 18709938
- [Background] Shafi S, Kauder DR. Fluid resuscitation and blood replacement in patients with polytrauma. Clin Orthop Relat Res. 2004 May;(422):37-42. doi: 10.1097/01.blo.0000129149.15141.0c. PMID 15187831
- [Derived] Akbuga Ozel B, Ozel G, Mamak Ekinci EB, Demirtola AE, Sahin G, Aksoy G, Yanikyurek I, Karaaslan MU. The MAR method versus the visual estimation method in predicting external blood loss: a randomized controlled study. Sci Rep. 2025 Aug 24;15(1):31091. doi: 10.1038/s41598-025-16169-0. PMID 40851079
- See also: Merlin MA, Alter SM, Raffel B, Pryor PW 2nd. External blood loss estimation using the MAR Method. Am J Emerg Med. 2009 Nov;27(9):1085-90. — https://pubmed.ncbi.nlm.nih.gov/19931755/